CLINICAL TRIAL: NCT06522126
Title: The Effects of Progressive Relaxation Exercise on Life Satisfaction, Anxiety, and Psychological Well-being in Students Experiencing Premenstrual Syndrome: A Randomized Controlled Trial
Brief Title: The Effects of Progressive Relaxation Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Esra SABANCI BARANSEL, Assistant professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022/3734
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Effects of Progressive Relaxation Exercise; Exercise; Relation, Interpersonal
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effects of progressive relaxation exercise (Experimental): Progressive relaxation exercises were given to female students who scored 111 and above on the PMS scale and were selected by randomization for the exercise group. The exercises were applied to those who participated in the study, met the inclusion criteria, and were able to participate in the study for 8 weeks. In the study, progressive relaxation exercises were applied by the researcher to the students in the exercise group with PMS complaints in the first three days of their first menstrual cycle.
  Interventions: Behavioral: progressive relaxation exercise
- control groups (No Intervention): Control group standard care group

INTERVENTIONS:
Behavioral: progressive relaxation exercise — One of the techniques employed to mitigate the prevalence of PMS complaints in women during this period is progressive relaxation exercises (PRE). It is one of the most preferred options due to its simplicity, cost-effectiveness, and reliability. Over the course of numerous years of research, progressive relaxation has been validated as an efficacious approach for regulating muscle tension. These exercises are performed to facilitate the distinction between tension and looseness in the body and to enable the individual to relax on her own in daily life. PRE involves the voluntary, systematic tension and relaxation of large muscle groups in the human body. PRE reduces anxiety levels by reducing muscle tension. It also provides the individual with a sense of profound rest, renewal, and rebirth.
  Arms: effects of progressive relaxation exercise

SUMMARY:
Aim: This research was conducted to determine the effects of progressive relaxation exercise on life satisfaction, anxiety, and psychological well-being in people experiencing premenstrual syndrome.

Methods: This randomized controlled trial was conducted with students who were enrolled in a university in the east of Türkiye, studying at the undergraduate levels outside the field of health, and experiencing premenstrual syndrome. The sample of the research consisted of 162 students (Exercise group 81 participants; Control group 81 participants). The Personal Information Form, Premenstrual Syndrome Scale (PMSS), Life Satisfaction Scale (LSS), Beck Anxiety Scale (BAS), and Psychological Well-Being Scale (PWBS) were used to collect data. Women in the exercise group underwent eight sessions of relaxation exercises, once a week for 8 weeks. In addition, for eight weeks after the first exercise, the participants exercised at home, at least twice a week, outside of the training. The PMSS, LSS, BAS, and PWBS were applied as post-tests to the participants in both groups, 8 weeks after the pre-tests.

ELIGIBILITY:
Inclusion Criteria:

* Those who scored 111 points or more on the Premenstrual Syndrome Scale,
* were married or single at the time of the research,
* did not have children.

Exclusion Criteria:

* those who were pregnant or postpartum,
* those who were diagnosed with any psychiatric disease according to the records,
* those who did not perform relaxation exercises outside of the training.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 162 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | 8 weeks
  It is a 44-item Likert-type scale developed by Gençdoğan (2006) that measures the severity of premenstrual symptoms. The scale has nine subscales, and the "PMSS total score" consisting of the scores related to the subscales and the total of the scale is obtained. The application of PMSS is done by retrospectively evaluating the person's status "one week before menstruation". The lowest score that can be obtained from the scale is 44 and the highest score is 220. The higher the score, the more intense the premenstrual syndrome symptoms are considered. The highest score that can be obtained for the total score is 220, 50% of which is 110 points. Therefore, those who score 111 and higher have PMS in terms of total score.

SECONDARY OUTCOMES:
Life Satisfaction Scale (LSS) | 8 weeks
  The scale was developed by Diener et al. Cronbach's alpha reliability coefficient of the scale was determined

OTHER OUTCOMES:
Beck Anxiety Scale (BAS) | 8 weeks
  The scale was developed by Beck et al. to determine the incidence of anxiety and anxiety symptoms experienced by individuals. The scoring of the measurement, which consists of 21 items, varies between 0-3. The scale was adapted into Turkish by Ulusoy et al. As a result of studies conducted with individuals presenting with psychological complaints

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Sabanci Baransel, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No individual participant data were not shared